CLINICAL TRIAL: NCT00782756
Title: A Phase II Study of Bevacizumab, Temozolomide and Hypofractionated Radiotherapy for Patients With Newly Diagnosed Malignant Glioma
Brief Title: Bevacizumab, Temozolomide and Hypofractionated Radiotherapy for Patients With Newly Diagnosed Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-126
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2017-03

CONDITIONS: Brain Cancer; Malignant Glioma
Keywords: Radiation; BEVACIZUMAB; AVASTIN; TEMOZOLOMIDE; newly diagnosed; Glioblastoma; GBM; malignant glioma; Radiotherapy; 08-126
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma | interventions — Radiotherapy; Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- RT, with temozolomide and bevacizumab (Experimental): This treatment regimen is novel in that it delivers the initial course of RT over 2 weeks instead of 6 weeks; also, the addition of bevacizumab during and after RT is a new approach.
  Interventions: Other: radiotherapy (RT) in combination with temozolomide and bevacizumab

INTERVENTIONS:
Other: radiotherapy (RT) in combination with temozolomide and bevacizumab — Bevacizumab10 mg/kg IV once every two weeks on days 1 and 15 of every cycle (Cycle defined as 28 days). Temozolomide 75mg/m2 daily beginning on day 1 through completion of radiotherapy. Hypofractionated dose painting IMRT will start on day 1 and will be delivered on a Monday, Wednesday, Friday schedule for a total of 6 fractions.
  Post RT therapy: Bevacizumab 10mg/kg IV every two weeks. Temozolomide 150-200mg/m2 daily for 5 consecutive days will be given on 28 day cycles.
  Follow up: CBC weekly, comprehensive panel and urinalysis monthly, blood pressure every other week. Neurological/physical examination monthly. Gd-enhanced MRI with perfusion every 2 cycles. Neurocognitive testing (approximately 4months post RT, 1 year after diagnosis and then annually in long term survivors). Blood sample for correlative studies monthly.

SUMMARY:
The purpose of this study is to test the safety of a new plan for treating glioblastoma. The usual first treatment for glioblastoma is to give focused radiation over 6 weeks in combination with a chemotherapy called temozolomide. In this study the radiation will be given over 2 weeks in combination with temozolomide and another drug, bevacizumab, will also be given. Our idea is that this treatment plan may attack both the tumor and the blood vessels feeding the tumor more effectively. This study will look at what effects, good or bad, this approach has on the patient and the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of glioblastoma or grade IV glioma.
* Tumor volume should be less than 60 cc (approximately 5cm maximum diameter).
* Age > or = to 18
* KPS ≥70
* Granulocyte count >1.5 X 10 9/L
* Platelet count >99 X 10 9/L
* SGOT < 2.5X upper limit of normal (ULN)
* Serum creatinine < 2X ULN
* Bilirubin < 2X ULN
* All patients must sign written informed consent

Exclusion Criteria:

* Any prior chemotherapy, radiotherapy and biologic therapy for glioma.
* Any prior experimental therapy for glioma.
* Multicentric glioma
* Other concurrent active malignancy (with the exception of cervical carcinoma in situ or basal cell ca of the skin).
* Serious medical or psychiatric illness that would in the opinion of the investigator interfere with the prescribed treatment.
* Pregnant or breast feeding women.
* Refusal to use effective contraception
* Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 12 months prior to Day 1
* History of stroke or transient ischemic attack
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of treatment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a UPC ratio ≥ 1.0 at screening
* Known hypersensitivity to any component of bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10-28 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Omuro, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- RT, With Temozolomide and Bevacizumab: This treatment regimen is novel in that it delivers the initial course of RT over 2 weeks instead of 6 weeks; also, the addition of bevacizumab during and after RT is a new approach.
  Bevacizumab10 mg/kg IV once every two weeks on days 1 and 15 of every cycle (Cycle defined as 28 days). Temozolomide 75mg/m2 daily beginning on day 1 through completion of radiotherapy. Hypofractionated dose painting IMRT will start on day 1 and will be delivered on a Monday, Wednesday, Friday schedule for a total of 6 fractions.
Period: Overall Study
Arm/Group | RT, With Temozolomide and Bevacizumab
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RT, With Temozolomide and Bevacizumab
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 55 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Safety assessments and toxicity grading will follow CTCAE Version 4 Grade
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | RT, With Temozolomide and Bevacizumab
Number analyzed (Participants) | 40
Participants | 40

2. Secondary Outcome: Progression Free Survival
Time Frame: through study completion, an average of 1 year
Measure: Median (Full Range); unit: months
Arm/Group | RT, With Temozolomide and Bevacizumab
Number analyzed (Participants) | 40
months | 10 [8 to 11]

3. Secondary Outcome: Neurocognitive Outcome
Time Frame: through study completion, an average of 1 year
Population: 37 participants agreed to undergo neuropsychological evaluations.
Measure: Count of Participants; unit: Participants
Arm/Group | RT, With Temozolomide and Bevacizumab
Number analyzed (Participants) | 40
Participants
  Neuropsychological evaluations | 37
  Did not agree to neuropsychological evaluations | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | RT, With Temozolomide and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 40/40
Serious Adverse Events (participants affected / at risk) | 19/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RT, With Temozolomide and Bevacizumab (N=40)
Colitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 1
Creatinine (Investigations) | 2
Glomerular filtration rate (Renal and urinary disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Hemorrhage, CNS (Nervous system disorders) | 1
Infection, other (Infections and infestations) | 2
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Muscle weakness - Left-sided (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Ocular/Visual - Other (specify) (Eye disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Pain - Head/headache (Nervous system disorders) | 2
Personality/behavioral (Psychiatric disorders) | 1
Platelets (Investigations) | 6
Pyramidal tract dysfunction (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 13
Speech impairment (Nervous system disorders) | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 3
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 3
Vasovagal episode (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RT, With Temozolomide and Bevacizumab (N=40)
Fatigue (General disorders) | 29
Constipation (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 15
Headache (Nervous system disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 7
Diarrhea (Gastrointestinal disorders) | 6
Mucositis oral (Gastrointestinal disorders) | 12
Hemorrhage/Bleeding - other (Injury, poisoning and procedural complications) | 4
Hypertension (Vascular disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Leukocytes (total WBC) (Investigations) | 3
Neuropathy - sensory (Nervous system disorders) | 3
Pain - Joint (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Hemorrhage, Nose (Respiratory, thoracic and mediastinal disorders) | 2
Hemorrhage, Oral cavity (Gastrointestinal disorders) | 2
Memory Impairment (Nervous system disorders) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Pain - neck (Musculoskeletal and connective tissue disorders) | 2
Platelets (Investigations) | 2
Proteinuria (Renal and urinary disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Seizure (Nervous system disorders) | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 2
Vision-blurred vision (Eye disorders) | 2
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-04-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT00782756/Prot_SAP_000.pdf